CLINICAL TRIAL: NCT06814314
Title: Pilot Study of Transcriptomic Alterations Associated with Antipsychotic-induced Metabolic Disorders in Children and Adolescents
Brief Title: AP Metabolism Transcriptomics
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: 9/24 (ex 995)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Neurodevelopmental Disorders; Irritability
Keywords: antipsychotic drugs; dyslipidemia; pre-diabetes; obesity; transcriptomics
MeSH Terms: conditions — Neurodevelopmental Disorders; Dyslipidemias; Glucose Intolerance; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- AP+ / MetS+: Persons using antipsychotic drugs and meeting diagnostic criteria for the metabolic syndrome
  Interventions: Diagnostic Test: Transcriptomic investigation
- AP+ / MetS-: Persons using antipsychotic drugs not meeting diagnostic criteria for the metabolic syndrome
  Interventions: Diagnostic Test: Transcriptomic investigation
- AP- / MetS+: Persons meeting diagnostic criteria for the metabolic syndrome not using antipsychotic drugs
  Interventions: Diagnostic Test: Transcriptomic investigation

INTERVENTIONS:
Diagnostic Test: Transcriptomic investigation — Transcriptomic investigation followed by ontology classification

SUMMARY:
It is known from the literature that treatment with antipsychotic drugs (AP) induces, even before changes in blood chemistry parameters, changes in gene transcription that are evident at the level of peripheral blood mononuclear cells.

In this pilot study we intend to evaluate the transcriptomic profile of children and adolescents who are undergoing treatment with antipsychotics and show metabolic disorders, in order to compare it to the profile of similar patients who do not use antipsychotics, but show metabolic disorders, or who use antipsychotics, but do not show metabolic disorders.

The hypothesis is that a different transcriptomic profile can be identified between the three populations under study, such as to allow to hypothesize that a series of transcripts can be used as early biomarkers of whether treatment with antipsychotics can induce metabolic disorders in the individual patient or not. This information could be used to improve the management of antipsychotic therapies in the direction of personalized medicine, reducing metabolic risks.

ELIGIBILITY:
Inclusion Criteria:

* age 5-17 years;
* group 1: antipsychotic users with metabolic disorders;
* group 2: antipsychotic users without metabolic disorders;
* group 3: non-antipsychotic users with metabolic disorders. The definition of antipsychotic use includes daily use for at least 3 months prior to enrollment.

The definition of metabolic disorders includes: BMI-Z for age, sex and height > +1 Waist circumference > 90th percentile for age, sex and height Diastolic or systolic blood pressure > 90th percentile for age, sex and height Fasting blood glucose > 99 mg/dl Fasting triglycerides > 149 mg/dl Fasting cholesterol < 41 mg/dl.

Patients with metabolic disorders are defined as those who meet at least one of the above criteria.

Patients without metabolic disorders are defined as those who do not present any of the above criteria.

Exclusion Criteria:

* presence of diagnosed genetic conditions known to alter energy metabolism and/or nutrition;
* presence of diagnosed eating disorders;
* habitual use of supplements known to alter energy metabolism and/or nutrition;
* concomitant use of drugs known to alter energy metabolism and/or nutrition.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Persons with metabolic syndrome and/or users of antipsychotic drugs
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
BMI-Z | Once, at recruitment
  Body mass index, normalized by age and sex. Values below -1 indicate underweight, values below 1 indicate overweight.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Eugenio Medea, Bosisio Parini, LC, Italy